CLINICAL TRIAL: NCT02841696
Title: Predictive Factors of Systolic Dysfunction in Non-complicated Hypertensive Patients (GLS OBservationAL Study in HyperTensioN - GLOBAL-HTN)
Brief Title: Predictive Factors of Systolic Dysfunction in Non-complicated Hypertensive Patients
Acronym: GLOBAL-HTN
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2014/07
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2016-07

CONDITIONS: Hypertension
Keywords: Heart failure; Systolic dysfunction; GLS; Arterial stiffness; Left ventricular hypertrophy
MeSH Terms: conditions — Hypertension; Heart Failure; Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hypertensive people: Hypertensive people recruited 10 years ago before any anti-hypertensive treatment
  Interventions: Device: Cardiac echography

INTERVENTIONS:
Device: Cardiac echography — The exam is in the left lateral decubitus position. 4 electrodes are applied to the patient's chest for a synchronization with the Electrocardiogram (ECG). The examination is conducted as standard with acquisition loops of records in parasternal long axis parasternal short axis, apical 4-cavities, 2-cavities and aorta 2 cavities.

SUMMARY:
Hypertension is a major cardiovascular risk factor. Heart failure is one of its main complications but the factors that influence its development are still insufficiently known. The primary objective is to determine associated factors to the occurrence of left ventricular (LV) systolic dysfunction assessed by an alteration of the Global Longitudinal Strain (GLS) after more than the years of hypertension. The secondary objective is to estimate the prevalence of LV systolic dysfunction in a cohort of hypertensive people followed for over 10 years and formulate pathophysiological hypotheses on the development of this heart disease.

DETAILED DESCRIPTION:
Some of the hypertensive patients will develop a post hypertensive heart disease. This hypertrophic cardiomyopathy is now essentially defined by the association of LV hypertrophy and diastolic dysfunction. Investigators believe this hypertrophic cardiomyopathy is also characterized by early impairment of systolic function but mainly in its longitudinal component (assessed by measuring the GLS) and therefore exposed to cardiovascular events.

The work is based on an existing cohort of hypertensive patients included more than 10 years ago before any initiation of antihypertensive therapy in the hypertension unit of the Bordeaux University Hospital, France. Patients will be contacted for further consultation with a cardiologist to identify patients with a LV systolic dysfunction. The primary end-point is a decrease of the longitudinal systolic function with a GLS<-17% for men and <-19% for women.

A sufficient number of patients will be contacted in order to collect data of at least 400 patients after more than 10-year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient who was diagnosed as hypertensive more than 10 years ago and who underwent cardiac-echography, ECG, a biological blood test and an ambulatory blood pressure measurement before the introduction of antihypertensive treatment.

Exclusion Criteria:

* Oral refusal of patient participation or its legal representatives, reading the specific information note for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject with a confirmed hypertension before any anti-hypertensive treatment more than 10 years ago.
  Patients are selected according their date of inclusion in the cohort. The investigators will start to contact the most recently recruited patients.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Measure of GLS | Day 1
  GLS measurement is a percentage obtained on cuts apical 4-chamber, 2-aortic cavities and 2 cavities (average of 3 impacts) after locating the aortic pulsed Doppler of the opening and closing of the aortic valve.
  GLS < -17% for men and < -19% for women.

CONTACTS AND LOCATIONS:
Overall Officials: Paul PEREZ, MD, Study Chair — University Hospital, Bordeaux
Locations (1):
- University Hospital Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No